CLINICAL TRIAL: NCT00982943
Title: The Epidemiological Study on Psychiatric Disorders and Psychotropic Drugs
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: I-Chih Cheng, Department of Psychiatry
Other Study IDs: FEMH-97-C-022
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Last update posted 2009-09-23 (Estimated); Status verified 2009-09

CONDITIONS: Psychiatric Disorders
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
During the past decade, the dramatic change in patterns of both psychiatric diagnoses and prescription of psychotropic agents has been noted since the introduction of newer antidepressant drugs. In the meantime, suicide has been recognized as a major public health problem all over the world. Research efforts have hence been spent in exploring the interrelationships between suicide rates and prescription of antidepressant drugs (as a proxy for the treatment of depression). However, most available studies came from developed countries despite that the majority of countries with rising suicide rates during the past decade were developing countries. Both suicide rates and prescription of antidepressant agents have been rising in Taiwan during the past decade; with a reliable mortality registrar and nationwide health insurance covering 99% of its population, Taiwan is distinctive in realizing a large-scale analysis on these interrelationships between suicide and prescription of antidepressant drugs. However, there has been no study in Taiwan exploring these potential associations up to now.

This study aims at examining the interrelationships between suicide rates and prescription of antidepressant agents based on the health insurance data from persons who had diagnoses of ICD: 290-319 or were prescribed with antidepressant agents during the period from 1998 to 2006. The investigators plan to first perform correlation analyses between the trends of suicide rates and prescription of antidepressants during the study period after taking into accounts potential confounding factors; analyses by age, gender groups and by administrative regions will also be performed. Besides, the investigators plan to analyze the change in the prescription pattern of psychotropic agents in Taiwan during the study period, with the particular focus on that of newer antidepressant drugs. The prescription of psychotropic agents in both psychiatric and non-psychiatric diagnoses will be explored.

ELIGIBILITY:
Inclusion Criteria:

* psychiatric disorders

Exclusion Criteria:

* without psychiatric disorders

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: the health insurance data from persons who had diagnoses of ICD: 290-319 or were prescribed with antidepressant agents during the period from 1998 to 2006
Sampling Method: Probability Sample
Enrollment: 1000000 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, Taipei County, Taiwan